CLINICAL TRIAL: NCT04658758
Title: Risk Assessment and Incidence of Vein Infusion Phlebitis After Intravenous Infusion of Proton Pump Inhibitors
Brief Title: The Incidence and Risk of Vein Infusion Phlebitis After Intravenous Infusion of Proton Pump Inhibitors
Acronym: VeinIPP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201085; 2020-A02319-30 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-11-30; First posted 2020-12-08 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Vein Infusion Phlebitis
Keywords: vein infusion phlebitis; proton pump inhibitor therapy; intravenous infusion; ulcer bleeding; aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intermittent or continuous proton pump inhibitor (PPI) therapy are recommended for high-risk bleeding ulcers according to the French Society of Gastroenterology. The prevalence of incidence of vein infusion phlebitis after PPI intravenous infusion is high in geriatric acute ward (about 10% of severe vein infusion phlebitis).

The primary of objective of the study is to determinate the prevalence of vein infusion phlebitis after PPI intravenous infusion in aging people.

The secondary of objective of the study if to determinate the factors of risk of vein infusion phlebitis.

DETAILED DESCRIPTION:
This is a multicenter observational study. 5 centers will participate to the study. Aging patients undergoing PPI intravenous infusion therapy will be proposed to be enrolled in the study. Paramedical observation will be performed during 5 days for each enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 70 years;
* Undergo intravenous continuous or intermittent proton pump inhibitor therapy;
* Patients being informed and not opposed to the study.

Exclusion Criteria:

* Existing vein infusion phlebitis before the PPI infusion by intravenous route;
* Under guardianship or curators;
* Covered by french AME health system.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patients aged > 70 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Occurence of infusion phlebitis | at day-5
  The Visual Infusion Phlebitis Scale will be used to define.

SECONDARY OUTCOMES:
Factors of risk of vein infusion phlebitis | Throughout of the study, an average of 1 year
  To determinate risk factors for vein infusion phlebitis.

CONTACTS AND LOCATIONS:
Overall Officials: Marion PEPIN, MD, PhD, Principal Investigator — Geriatric Department, Ambroise Paré Hospital, APHP
Locations (1):
- Geriatric Department, Ambroise Paré Hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No